CLINICAL TRIAL: NCT07036380
Title: MP0317, a Tumor Targeting FAP Dependent CD40 Agonist DARPin, in Combination With Chemoimmunotherapy in First Line Treatment for Patients With Advanced Biliary Tract Carcinoma: a Radnomized Non-comparative Proof of Concept Phase II Study
Brief Title: MP0317 in Combination With Chemoimmunotherapy in First Line Treatment for Patients With Advanced Biliary Tract Carcinoma
Acronym: TACTIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/926; 2024-520029-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-15; First posted 2025-06-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Advanced Biliary Tract Carcinoma
Keywords: immunotherapy; DARPin; Advanced Biliary Tract Carcinoma
MeSH Terms: interventions — Gemcitabine; durvalumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MP0317 + Gemcitabine + Cisplatin + Durvalumab (Experimental): MP0317- Gemcitabine+ Cisplatin + Durvalumab
  Interventions: Drug: MP0317 + Gemcitabine + Cisplatine + Durvalumab; Procedure: CT-Scan
- Gemcitabine + Cisplatin + Durvalumab (Active Comparator): Gemcitabine + Cisplatin + Durvalumab
  Interventions: Procedure: CT-Scan; Drug: Gemcitabine + Cisplatin + Durvalumab

INTERVENTIONS:
Drug: MP0317 + Gemcitabine + Cisplatine + Durvalumab — * MP0317: 3 mg/kg IV(intraveinous), day 1, every 3 weeks for a maximum of 5 administrations
  * Immuno-chemotherapy (ICT): cycle 1-5
    * Durvalumab 1500 mg IV, day 8 every 3 weeks
    * Gemcitabine 1000 mg/m² IV, days 8 and 15 every 3 weeks
    * Cisplatin 25 mg/m² IV, days 8 and 15 every 3 weeks
  * Immuno-chemotherapy (ICT): cycle 6-8
    * Durvalumab 1500 mg IV every 3 weeks
    * Gemcitabine 1000 mg/m² at day 1, 8 every 21 days
    * Cisplatin 25 mg/m² at day 1, 8 every 21 days
  * Then durvalumab (1500 mg IV) will be administrated in monotherapy maintenance every 4 weeks until progression or unacceptable toxicity.
  Arms: MP0317 + Gemcitabine + Cisplatin + Durvalumab
Procedure: CT-Scan — at baseline, every 6 weeks (± 1 week) for the first 24 weeks and then every 8 weeks until progression, at end of treatment visit, At each follow-up visit : Only for patients who have not progressed during treatment phase
Drug: Gemcitabine + Cisplatin + Durvalumab — * Immuno-chemotherapy (ICT) for 8 cycles :
    * Durvalumab 1500 mg IV, day 1 every 3 weeks
    * Gemcitabine 1000 mg/m² IV, days 1 and 8 every 3 weeks
    * Cisplatin 25 mg/m² IV, days 1 and 8 every 3 weeks
  * Then durvalumab (1500 mg IV) will be administrated in monotherapy maintenance every 4 weeks until progression or unacceptable toxicity.
  Arms: Gemcitabine + Cisplatin + Durvalumab

SUMMARY:
In the present TACTIC clinical trial, the investigators propose to determine the clinical interest and immunological efficacy of a treatment combining MP0317 the FAP (Fibroblast Activation Protein)-dependent CD40 agonist, with anti-PD-L1(Programmed Death-Ligand 1) therapy (durvalumab) and gemcitabine-cisplatin-based chemotherapy in unresectable cholangiocarcinoma.

The main objective is to assess the 12-month progression free survival (PFS) rate in the experimental arm. The trial proposed is a non-comparative proof of concept randomized two-stage phase II. The control arm will serve to verify the good calibration of the null hypothesis made in the experimental arm and to provide "true" controls for translational investigations. A semi-continuous monitoring of toxicity is planned in the experimental arm during the first stage of the study to warrant the tolerability of the experimental treatment and then to guarantee the security of the patients.

75 patients (50 in the experimental arm) will be included. The investigators will also decipher, as a translational objective, the molecular and immunological parameters determining the clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent
2. Histologically confirmed biliary tract carcinoma: intra/extrahepatic cholangiocarcinoma (note that gallbladder carcinoma are not eligible)
3. Locally advanced unresectable or metastatic
4. Patient who had not previously received systemic anti-cancer treatment (adjuvant treatment with Capecitabine is allowed if the end of the chemotherapy was at least 6 months ago)
5. Age ≥ 18 years
6. Measurable disease defined according to RECIST v1.1 (Response Evaluation Criteria In Solid Tumours) guidelines Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.
7. Patients who have received previous chemoembolization, radioembolization and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 according to National Cancer Institute [NCI] common terminology criteria for adverse events, version 5 (CTCAE v5); with the exception of Grade 2 alopecia
8. Performance status ECOG-PS < 2 (Eastern Cooperative Oncology Group)
9. Females must be using highly effective contraceptive measures, and have a negative pregnancy test prior to the start of dosing if of childbearing potential, and during treatment and at least 7 months after the end of the treatment with cisplatin, 6 months after the end of the treatment with gemcitabine, 3 months after the end of the treatment with durvalumab, or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

   1. Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution.
   3. Women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
   4. Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and at least: 4 months after the end of the treatment with cisplatin and 3 months after the end of the treatment with gemcitabine. Patients should refrain from donating sperm from the start of dosing until 4 months after discontinuing study treatment.
10. Documented virology status of hepatitis, as confirmed by screening HBV and HCV tests:

    1. For patients with active HBV: HBV DNA <500 IU/ml (International unit)during screening, initiation of anti-HBV treatment at least 14 days prior to randomization and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir)
    2. Patients with HCV, either with resolved infection (as evidenced by detectable antibody) or chronic infection (as evidence by detectable HCV RNA), are eligible
11. Patient affiliated to or beneficiary of French social security system
12. Ability to comply with the study protocol, in the Investigator's judgment.

Exclusion Criteria:

For patients whose tumors present a genetic alteration of IDH1, FGFR2 or BRAF as well as an amplification of HER2, the investigators of the TACTIC study recommend, if possible, the orientation for preferential inclusion in the SAFIR ABC10 study".

1. Patients previously exposed to anti-tumor immunotherapy such as anti-PD-1, anti-PD-L1, or anti-CTLA4 (cytotoxic T-lymphocyte-associated protein 4) agent or any immune therapy
2. Diagnosis of additional malignancy within 3 years prior to the inclusion with the exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer
3. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
4. Current participation in a study of an investigational agent or in the period of exclusion
5. Patient under guardianship, curatorship or under the protection of justice
6. Other liver malignancy: hepatocellular carcinoma and hepato-cholangiocarcinoma
7. Uncontrolled pleural effusion, pericardial effusion, ascites or symptomatic fistula
8. Uncontrolled tumor-related pain: exposing patients to risk of exposure to corticoids or iterative hospitalizations. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to inclusion. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
9. Known active central nervous system metastases and/or carcinomatous meningitis.
10. History of angiocholitis, liver abscess, or acute pancreatitis within 4 weeks prior to initiation of study treatment
11. Inadequate organ functions: known cardiac failure of unstable coronaropathy, respiratory failure, or uncontrolled infection or another life-risk condition. Patients requiring oxygen therapy or with LEVF<40% (Left ventricular ejection fraction).
12. HIV (human immunodeficiency virus) positive (HIV 1/2 antibodies patients), or a known history of active Tuberculosis bacillus
13. Any immunosuppressive therapy (i.e. corticosteroids >10 mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy
14. Active autoimmune disease that has required a systemic treatment in the past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    1. Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study
    2. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
    3. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

       * Rash must cover < 10% of body surface area,
       * Disease is well controlled at baseline and requires only low-potency topical corticosteroids,
       * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months,
15. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
16. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
17. Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of durvalumab
18. Receipt of a live, attenuated vaccine within 30 days prior to inclusion or anticipation that such a live, attenuated vaccine will be required during the study Note: Patients must agree not to receive live, attenuated influenza vaccine within 28 days prior to randomization, during treatment or within 5 months following the last dose of durvalumab
19. Inadequate hematology function: Lymphocyte count at baseline < 700/mm3; neutrophil count < 1 500/mm3, platelets < 10 0000/mm3 (without transfusion), Hemoglobin < 9g/dL (patients may be transfused to meet this criterion).
20. Inadequate hepatic function: bilirubin >2 fold ULN (upper limit of normal), AST/ALT >3 fold ULN, International normalized thromboplastin time ratio >2
21. Creatinine clearance (CrCl) < 60 ml/min (by the Modification of Diet in Renal Disease [MDRD], Cockroft formula, or chronic kidney disease [CKD] formula])
22. Serum albumin < 28 g/L
23. Surgery within 4 weeks previously the initiation of the study treatment
24. Radiotherapy within 2 weeks previously the initiation of the study treatment
25. Patient with weight < 36 kg.
26. Pregnant or breastfeeding woman
27. Known hypersensitivity to components of MP0317, for exemple, histidine buffer or the Tween diluent, according to section 7.2 " Contraindications " of the Investigator's brochure of MP0317
28. Hypersensitivity to gemcitabine or to cisplatin, or to any of their excipients, according to the SmPCs of these products
29. According to the SmPC of cisplatin: hearing problem, in case of combination with phenytoin with prophylactic aim, patients with neuropathy caused by cisplatin, in case of cardiorespiratory pathology in particular, which forbids a hyperhydration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
progression free survival status (PFS) at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BORG, Study Director — CHU Besançon
Locations (11):
- France (11):
  - CHU de Besançon, Besançon
  - Centre georges-François Leclerc, Dijon
  - CHU de Grenoble, Grenoble
  - Centre Léon Bérard, Lyon
  - CHU de Montpellier, Montpellier
  - Hôpital Beaujon, Paris
  - Hôpital La Pitié-Salpétrière, Paris
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - CHU de Tours, Tours
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No